CLINICAL TRIAL: NCT06763601
Title: Effect of Shoulder Symptom Modification Procedure (SSMP) in Managing Patients with Frozen Shoulder: a Pilot Study
Brief Title: Effect of Shoulder Symptom Modification Procedure (SSMP) in Managing Patients with Frozen Shoulder
Acronym: SSMP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gulf Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-COHS-STD-112-Dec-2024; Internal review board (Other: Gulf medical University)
Record Dates: First submitted 2024-12-11; First posted 2025-01-08 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2024-12

CONDITIONS: Frozen Shoulder
Keywords: SSMP; MWM; sham mobilization; frozen shoulder
MeSH Terms: conditions — Bursitis | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: each participant will be randomly allocated one group. there are three groups in total
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- SSMP (Experimental): SSMP, Isometric exercise, eccentric exercise, heavy slow resistance , functional program
  Interventions: Procedure: SSMP, Isometric exercise, eccentric exercise, heavy slow resistance , functional program
- MWM (Experimental): MWM procedure followed by Isometric exercise, eccentric exercise, heavy slow resistance , functional program
  Interventions: Procedure: MWM,Isometric exercise, eccentric exercise, heavy slow resistance , functional program
- sham mobilization (Placebo Comparator): Sham mobilization will be given for placebo effect followed by Isometric exercise, eccentric exercise, heavy slow resistance , functional program
  Interventions: Procedure: sham mobilization

INTERVENTIONS:
Procedure: SSMP, Isometric exercise, eccentric exercise, heavy slow resistance , functional program — In this group the patients will be given symptom modification procedure in the first phase followed by isometric exercises in second phase, eccentrics and HSR in third phase and functional program in fourth phase
  Arms: SSMP
Procedure: MWM,Isometric exercise, eccentric exercise, heavy slow resistance , functional program — in this mobilization with movement in first phase will be given followed by isometrics, eccentrics and heavy slow resistance exercise and finally the functional program
  Arms: MWM
Procedure: sham mobilization — Sham mobilization followed by isometrics, eccentric training and heavy resistance training and finally the functional program .
  Arms: sham mobilization

SUMMARY:
the study is about intervention to patient with frozen shoulder to help patients improve function and shoulder disability , reduce pain and improve range of motion, the main aim of this study is to find out which treatment intervention SSMP , MWM and sham mobilization give effective results

ELIGIBILITY:
Inclusion Criteria:

* • Diagnosis of adhesive capsulitis confirmed by a healthcare professional.

  * Scores more than 2 in adhesive capsulitis scale
  * Range of motion affected in capsular pattern
  * Age between 40-65 years.
  * Willingness to participate by signing informed consent

Exclusion Criteria:

* Having any history of shoulder dislocation
* Humerus fractures or trauma
* Diagnosed with any sort of cancer
* History of cardiovascular disease

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-03-22 (Estimated); Study Completion 2025-05-16 (Estimated)

PRIMARY OUTCOMES:
Shoulder Pain And Disability Index | from enrollment to week 4,6,8
  shoulder pain and disability index is use to measure shoulder pain and disability where 0 is the best score and 130 is the worst
Numeric Pain Rating Scale | from enrollment to 8 weeks
  numeric pain rating scale where 0 indicates no pain and 10 indicates worst pain

SECONDARY OUTCOMES:
Range Of Motion | week 4,6,8
  range of motion of shoulder joint that includes flexion, extension abduction, adduction, internal and external rotation
Patients' Global Impression of Change (PGIC) scale | at enrollment and on 8th week
  PGIC is a 7 point scale depicting a patient's rating of overall improvement. where 1 indicates very much improved and 7 indicates worst

CONTACTS AND LOCATIONS:
Locations (1):
- Thumbay Physical Therapy and Rehabilitation Hospital, Ajman, United Arab Emirates

IPD SHARING:
Plan to Share IPD: Undecided